CLINICAL TRIAL: NCT06787846
Title: EVALUATION of the EFFICACY and TOLERABILITY of TESTED FORMULA VS. HYDROQUINONE 4% in the TREATMENT of FACIAL MELASMA OVER 3 MONTHS
Brief Title: EFFICACY and TOLERABILITY of TESTED FORMULA VS. HYDROQUINONE 4% in the TREATMENT of FACIAL MELASMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21028 - Serum vs HQ4%
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Melasma
Keywords: Melasma; Hydroquinone
MeSH Terms: conditions — Melanosis | interventions — hydroquinone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group TP: Tested product (Experimental): Subjects (aged over 18 years) with mild to severe facial epidermal or mixed melasma
  Interventions: Other: Experimental: Group TP
- Group HQ: Hydroquinone 4% (Active Comparator): Subjects (aged over 18 years) with mild to severe facial epidermal or mixed melasma
  Interventions: Drug: Active Comparator: Group HQ: Hydroquinone 4%

INTERVENTIONS:
Other: Experimental: Group TP — Serum : Application full face, twice daily, in the morning and at bedtime for 4 months and application Tinted sunscreen SPF 50+, twice a day
  Other Names: Tested Product
  Arms: Group TP: Tested product
Drug: Active Comparator: Group HQ: Hydroquinone 4% — Cream : Application all over the face once a day (at bedtime) and Tinted sunscreen SPF 50+, twice a day
  Other Names: Hydroquinone
  Arms: Group HQ: Hydroquinone 4%

SUMMARY:
This study aims at assessing the non-inferiority of tested formula facial serum (2039125 03) versus hydroquinone 4% over 3 months for treatment and then 3 months for maintenance ofwomen subjects presenting facial melasma.

DETAILED DESCRIPTION:
Topical treatments are usually used first line. Among a high number of molecules claiming a depigmenting effect, hydroquinone used at various concentrations (typically 2 to 5%) is the most widely used skin depigmenting product and is considered, up to now, the gold standard when used at 4-5%.

Hydroquinone is sometimes combined in the Kligman's trio, with topical tretinoin and topical steroids, which remains the best initial treatment for melasma in terms of efficacy.

This randomized , two-arm study is carried out with a new cosmetic formulation developed with the aim of acting on facial hyperpigmentation.

This clinical trial is conducted in accordance with the protocol, the HELSINKI declaration (1964) and subsequent amendments, and/or the International Council on Harmonization (ICH) Good Clinical Practices (GCP)/ and in compliance with applicable regulatory requirements.

Statistical Analysis:

* Primary Efficacy Analysis: The primary performance endpoint is the difference between tested formula facial serum (2039125 03) versus hydroquinone 4% in mean change from baseline in modified Melasma Area Severity Index (mMASI) score at D84. A non-inferiority followed by a superiority evaluation will be assessed.
* Sensitivity analyses The same analysis will be repeated on the FAS population. Missing values (i.e. data of patients who dropped out the study or with no evaluable data) will not be imputed for this analysis.

Depending on the results of the baseline characteristics description, other sensitivity analyses could be performed by adding other relevant baseline covariables to the model.

. Safety Analysis: no statistical analysis will be performed on safety. The data are presented descriptively.

Categorical data are summarized using the number and percentage of patients in each category. Continuous data are summarized using the arithmetic mean, Standard Deviation (SD), Q1, Q3, minimum, median and maximum values.

Regarding the sample size determination, there was no formal calculation. A number of 104 patients , 52 patients in each group was considered sufficient to meet the study objective.

ELIGIBILITY:
Inclusion Criteria:

1. Women;
2. Adults (over 18 y.o.) (preference 18-50 y.o.);
3. Phototypes I to IV;
4. Melasma epidermal or mixed (exclude dermal melasma);
5. Ready to protect as much as possible from the sun for the duration of the study;
6. Ready to avoid contraindicated products (irritants, other depigmenting agents);
7. Participants demonstrating understanding of the study procedures, restrictions, and willingness to participate as evidenced by voluntary written informed consent and having received a signed and dated copy of the informed consent form.

Exclusion criteria

1. Subjects with dermal melasma (wood lamp at inclusion);
2. Subjects who has already use of hydroquinone 4% in the past year;
3. Subjects with stable hormonal therapy (contraceptive ou THS) for at least 6 months;
4. Pregnant or breastfeeding women or pregnancy plans;
5. Subjects applying irritants (such as peeling, acid..) (2 weeks wash out);
6. Subjects under active treatment of melasma (including topicals or procedures) within the last 2 weeks;
7. Subjects using drugs that can induce melasma such as antiepileptics (1 month wash out);
8. Subjects using other products claiming a depigmenting activity (1 month wash out);
9. Subjects with other dermatosis of the face or known photosensitivity;
10. All types of topical treatment applied to the face (wash out of 2 weeks)
11. Subjects without any facial procedure planned during the course of the study
12. Subjects under phototherapy (1 month wash out)
13. Subjects hypersensitivity to the products of the study
14. Any history of significant dermatological/ophthalmological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes,) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction
15. Subjects currently using any medication, which in the opinion of the investigator, may affect the evaluation of the study product, or place the subject at undue risk.
16. Previous history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, cosmetics, or medication
17. Participation in another clinical study
18. Employee of the sponsor or the study site

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Change in mMASI scoring | From baseline to 3months
  The mMASI is calculated using 3 components: four regions of the face (forehead, right malar, left malar and chin); area of involvement for each region (using a scale from 0 to 6): darkness compared to the surrounding normal skin for each area (evaluated using a scale from 0 to 4).
Evaluation of Global Tolerance | From 1month to 3 months
  The investigator evaluates the tolerance using a 5-point skin reaction scale (0 represent No local intolerance ; 4 represent a Very severe signs or symptoms of intolerance)

SECONDARY OUTCOMES:
Change in Investigator's Global Assessment (IGA) | From baseline to3 months
  The investigator evaluates the severity of melasma using a 4-point scale (from 0 (cleared, almost cleared) to 3 (severe (markedly darker than the surrounding normal skin)).
Change in Subject Global Assessment of Improvement (SGAI) | From 1month to 3 months
  The subject evaluates the change on a 6-point scale from -1 (worsened) to 4 (totally cleared).
Change of Quality of life | From 1month to 3 months
  Subjects evaluate about the impact of melasma on the quality of life. On a scale of 1 (not bothered at all) to 7 (bothered all the time), the subject's rate how they feel. MELAS Qol scores range from 7 to 70, with a higher score signifying worse quality of life.
Change of stigmatization evaluation | From 1month to 3 months
  Subjects evaluate about the impact of melasma on stigmatization evaluation. On a scale of 1 (not bothered at all) to 7 (bothered all the time), the subject's rate how they feel. MELAS Qol scores range from 7 to 70, with a higher score signifying worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Moura, Principal Investigator — CIDP
Locations (1):
- CIDP, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Passeron T, Kerob D, Le Dantec G, Demessant-Flavigny AL, do Nascimento AR, Moura R, Salah S, Feiges M, Fernandez E, Alexis A. Efficacy and Tolerability of a New Facial 2-Mercaptonicotinoyl Glycine-Containing Depigmenting Serum Versus Hydroquinone 4% over 3-Month Treatment of Facial Melasma. Dermatol Ther (Heidelb). 2025 Sep;15(9):2379-2390. doi: 10.1007/s13555-025-01473-4. Epub 2025 Jun 30. PMID 40586974